CLINICAL TRIAL: NCT02883543
Title: Phase III Study of Icotinib With Concurrent Radiotherapy as First-line Treatment for Unresectable/Oligometastasis NSCLC With EGFR Activating Mutation: a Prospective, Multicentre, Open-label, Randomised Study
Brief Title: First-line Icotinib With Concurrent Radiotherapy for NSCLC With EGFR Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhen-zhou Yang, Director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RILI2016
Record Dates: First submitted 2016-08-08; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- icotinib plus radiotherapy (Experimental): Eligible patients are administered with oral icotinib 125mg three times daily for two months, in which responsive patients (partial response and stable disease) are randomized (1: 1: 1) and receive icotinib plus concurrent radiotherapy.
  Interventions: Drug: icotinib; Radiation: Radiotherapy
- icotinib (Active Comparator): Eligible patients are administered with oral icotinib 125mg three times daily for two months, in which responsive patients (partial response and stable disease) are randomized (1: 1: 1) and receive icotinib monotherapy.
  Interventions: Drug: icotinib
- chemotherapy plus radiotherapy (Active Comparator): Eligible patients are administered with oral icotinib 125mg three times daily for two months, in which responsive patients (partial response and stable disease) are randomized (1: 1: 1) and receive chemotherapy plus concurrent radiotherapy.
  Interventions: Drug: Chemotherapy; Radiation: Radiotherapy

INTERVENTIONS:
Drug: icotinib — Icotinib is orally administered three times per day.
  Arms: icotinib; icotinib plus radiotherapy
Drug: Chemotherapy — Chemotherapy is given by intravenous administration. Three regimens are available in this study.
  Regimen 1: etoposide 75mg/m2 d1-5 + cisplatin 75 mg/m2 day1/ day1-2.
  Regimen 2: docetaxel 75mg/m2 d1 + cisplatin 75 mg/m2 day1/ day1-2.
  Regimen 3: pemetrexed 500mg/m2 d1 + cisplatin 75 mg/m2 day1/ day1-2
  Arms: chemotherapy plus radiotherapy
Radiation: Radiotherapy — 5Gy/75.00Gy, 10f/2w for peripheral lung cancer, and 2.4Gy/59.52Gy, 20f/4w for central lung cancer.
  Arms: chemotherapy plus radiotherapy; icotinib plus radiotherapy

SUMMARY:
Eligible patients are administered with oral icotinib 125mg three times daily for two months, in which responsive patients (partial response and stable disease) are randomized (1: 1: 1) and receive icotinib plus concurrent radiotherapy, or chemotherapy plus concurrent radiotherapy, or icotinib monotherapy.

DETAILED DESCRIPTION:
Eligible patients are administered with oral icotinib 125mg three times daily for two months, in which responsive patients (partial response and stable disease) are randomized (1: 1: 1) and receive icotinib plus concurrent radiotherapy, or chemotherapy plus concurrent radiotherapy, or icotinib monotherapy. The primary endpoint is progression-free survival, and the incidence of radiation-induced lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years
* Pathologically documented NSCLC
* Unresectable stage III or oligometastasis (less than three metastasis lesions, brain metastasis is not permitted) stage IV confirmed by CT and/or MRI
* Positive EGFR mutation confirmed by ARMS
* At least 3-month life expectancy
* KPS ≥ 70
* Adequate hematological values: hemoglobin ≥ 100 g/L, absolute neutrophils count ≥ 1.5 x 109/L, platelets count ≥ 100 x 109/L
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 1.5 x ULN
* Written informed consent before patient registration and any protocol-related procedures

Exclusion Criteria:

* Previous radiotherapy
* Received other investigational systemic drugs within 4 weeks prior to study entry
* Severe or uncontrolled systemic disease
* Active autoimmune disease, or a documented history of autoimmune/acquired immune disease, or a history of organ transplant
* Pregnant or lactating, women of childbearing potential, unless using effective contraception as determined by the investigator
* Any other serious underlying medical (e.g. active uncontrolled infection, active gastric ulcer, uncontrolled seizures), psychological and other condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
Incidence of radiation injure of the lungs | 2 years
  Measured according to NCI CTCAE v4.0

SECONDARY OUTCOMES:
Overall survival | 5 years
Tumor response after icotinib induction | 8 weeks
Quality of life | 2 years
  Measured by FACT-L

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhou Yang, MD, Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University

IPD SHARING:
Plan to Share IPD: No